CLINICAL TRIAL: NCT00460473
Title: A Phase III,Randomized, Double-Blind, Placebo-Controlled, Two-Arm Parallel, Multicenter Study Evaluating the Efficacy and Safety of Dexmedetomidine in the Prevention of Postoperative Delirium in Subjects Undergoing Surgery for Fractured Hip With General Anesthesia
Brief Title: A Research Study to Evaluate the Effectiveness of Dexmedetomidine in Preventing Delirium After Hip Fracture Repair Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The incidence of post-operative delirium observed from interim blinded data was significantly lower than the current literature in this population.
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DEX-06-09
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Delirium
Keywords: Mental Health; Neurological Disease; Hip Injuries and Disorders
MeSH Terms: conditions — Delirium; Psychological Well-Being; Nervous System Diseases; Hip Injuries; Disease | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Placebo (PBO) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine
  Arms: Dexmedetomidine
Drug: Placebo
  Arms: Placebo (PBO)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of perioperative use of dexmedetomidine in the prevention of postoperative delirium in subjects undergoing surgery for fractured hip with general anesthesia.

DETAILED DESCRIPTION:
Postoperative delirium is an acute decline in cognition and attention which is usually transient but when delirium persists it can impact cognitive function, morbidity and morality. There are no drugs that are currently approved to prevent the onset of delirium but dexmedetomidine has the potential to meet this unmet medical need. Hip fractures, unfortunately are frequent occurrences in the elderly population and the elderly are more prone to developing delirium after surgery.

Dexmedetomidine is currently approved for use for 24 hours in patients on ventilators in the ICU. Study participation will last from within 72 hours of surgery to 3 days after surgery, continue throughout surgery and up to 2 hours after surgery. Delirium will be assessed prior to surgery and for 72 hours after surgery. This assessment will consist of questions to determine memory and thought process. At discharge patient's resource utilization will be evaluated and thirty days after surgery questions will be asked regarding quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years old) male or female who will undergo surgery for fractured hip with general anesthesia within 72 hours of admission to hospital.
2. If female, subject is non-lactating and is either:

   1. Not of childbearing potential, defined as post-menopausal for at least 1 year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy or hysterectomy.
   2. Of childbearing potential but is not pregnant at time of baseline and is practicing one of the following methods of birth control: oral or parenteral contraceptives, double-barrier method, vasectomized partner, or abstinence from sexual intercourse.
3. Subject is American Society of Anesthesiologists Physical Status I, II, III, or IV.
4. Subject (or subject's legally authorized representative) has voluntarily signed and dated the informed consent document approved by the Institutional Review Board (IRB).

Exclusion Criteria:

1. Cognitive function level by Mini Mental State Exam (MMSE) of ≤20.
2. Subject has a positive CAM-ICU result for delirium at Screening or Baseline.
3. Subject requires chronic antipsychotic therapy.
4. Subject is anticipated to require additional surgical procedures during the 72 hour Screening Period and the 3 days Follow-up Period.
5. Subject is anticipated to require repair of pelvic fractures (eg,acetabulum).
6. Subject has participated in a trial with any experimental drug or experimental implantable device within 30 days prior to the study drug administration, or has ever been enrolled in this study.
7. Subject known to be in liver failure.
8. Subject has an anticipated potential for increased intracranial pressure or an uncontrolled seizure disorder or known psychiatric illness that could confound a normal response during study assessment.
9. Subject has received treatment with a α2-agonist or antagonist (within 14 days of study entry).
10. Subject for whom opiates, benzodiazepines, DEX or other α2-agonists are contraindicated.
11. Subject has, per the investigator's judgment, a known or suspected physical or psychological dependence on an abused drug, other than alcohol.
12. Subject has acute unstable angina, acute myocardial infarction, HR <50 bpm, SBP <90 mmHg, or third degree heart block unless the subject has a pacemaker.
13. Subject has any condition or factor which, in the Investigator's opinion, might increase the risk to the subject.
14. Subject is not expected to live more than 60 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who experienced any postoperative delirium up to 3 days after the end of study drug infusion | Twice daily (between 6:00-9:00 AM and 5:00-8:00 PM) until 3 days after the end of study drug infusion.
  The presence of postoperative delirium will be determined by Confusion Assessment Method for the Intensive Care Unit (CAM-ICU).

SECONDARY OUTCOMES:
Duration of postoperative delirium as determined by CAM-ICU up to 3 days after end of study drug infusion | Twice daily (between 6:00-9:00 AM and 5:00-8:00 PM) until 3 days after the end of study drug infusion.
Percentage of subjects who experienced postoperative delirium each day after end of study drug infusion | Twice daily (between 6:00-9:00 AM and 5:00-8:00 PM) until 3 days after the end of study drug infusion.
Perioperative use of all analgesics (Fentanyl, Morphine, and oral analgesics) | During the intraoperative period, Post-anesthesia care unit period and the 3 days Follow-up Period.
Postoperative use of Midazolam | During the PACU period (Approximately 2 hours)
  If RASS >0, midazolam (MDZ) 0.5-1 mg IV will be given until RASS <0. While in PACU during study drug infusion period, MDZ (0.5-1 mg IV) will be given if RASS >+1 under allowed maximum dose of study drug.
  RASS range:
  * +4 Combative -Overtly combative, violent, immediate danger to staff
  * +3 Very agitated- Pulls or removes tubes or catheters, aggressive
  * +2 Agitated- Frequent non-purposeful movements, fights ventilator
  * +1 Restless- Anxious, but movements not aggressive or vigorous
  * 0 Alert and calm
  * -1 Drowsy - Not fully alert, but sustained awakening (eye opening, eye contact) to voice (>10 sec)
  * -2 Light sedation - Briefly awakens with eye contact to voice (<10 sec)
  * -3 Moderate sedation - Movement or eye opening to voice (but no eye contact)
  * -4 Deep sedation No response to voice, but movement or eye opening to physical stimulation
  * -5 Unarousable No response to voice or physical stimulation
Time-to-Aldrete score of ≥9 | Every 15±5 minutes from arrival in the PACU (Approximately 2 hours)
  A score of 9-10 indicates the subject has recovered from anesthesia and is ready for discharge from the PACU.
Length of post-operative hospital stay | From the post operative period until subject discharged from hospital

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Loma Linda University Medical Center, Loma Linda, California
  - LAC-USC Medical Center Los Angeles, Los Angeles, California
  - Huntington Memorial Hospital, Pasadena, California
  - University of Miami-Jackson Memorial Medical Center, Miami, Florida
  - Southeastern Clinical Research Consultants, Orlando, Florida
  - Orlando Regional Healthcare, Critical Care Medicine, Orlando, Florida
  - G and G Research, Inc., Vero Beach, Florida
  - Orthopaedic Center of Vero Beach, Vero Beach, Florida
  - Medical College of Georgia, Augusta, Georgia
  - University of Iowa Hospitals and Clinics, Dept. of Anesthesia, Iowa City, Iowa
  - Outcomes Research Institute, Louisville, Kentucky
  - Louisiana State University, Dept. of Orthopaedic Surgery, Shreveport, Louisiana
  - Spectrum Health Blodgett Campus, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Saint Mary's Duluth Clinic Health System, Duluth, Minnesota
  - Mayo Clinic College of Medicine, Dept. of Anesthesiology, Rochester, Minnesota
  - University of Missouri, Columbia, Missouri
  - Mount Sinai School of Medicine, Great Neck, New York
  - New York University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Pittsburgh Medical Center, Presbyterian, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Research Concepts, Bellaire, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - University of Virginia Health Systems, Charlottesville, Virginia
  - University of Wisconsin Medical School, Dept. of Anesthesiology, Madison, Wisconsin
  - VA Medical Center, Milwaukee, Wisconsin